CLINICAL TRIAL: NCT01472874
Title: Single Daily Dosage of Trientine for Maintenance Treatment for Wilson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0902004694; ORPH-SYP-001 (Other: Valeant reference #)
Record Dates: First submitted 2011-11-11; First posted 2011-11-17 (Estimated); Results first posted 2014-05-19 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Wilson Disease
Keywords: Wilson Disease; Trientine; One Daily Dosage
MeSH Terms: conditions — Hepatolenticular Degeneration | interventions — Trientine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Once a day Trientine (Experimental): Patients receive once a day trientine
  Interventions: Drug: Once a day Trientine

INTERVENTIONS:
Drug: Once a day Trientine — Trientine at a dosage of ~15 mg/kg rounded upwards to the nearest 250 or 300 mg in a single daily dosage. The entire daily dosage will be taken at once in the AM an hour before any meal. Duration of the study is 1 year.
  Other Names: Syprine

SUMMARY:
Hypothesis: The investigators postulate that patients with Wilson disease who are asymptomatic or who have been effectively treated for their symptoms and are in a maintenance phase therapy can be safely and effectively treated with a single daily dosage of the chelating agent trientine.

Specific Aims: To demonstrate that a single daily treatment with trientine is as effective or better than a patient's current maintenance therapy. This will be accomplished by performance of a case control prospective study of patients on their prior therapy, and during a period of treatment with a single weight based dose regimen of trientine.

The primary endpoint for this study is the demonstration of equivalence to a patient's prior therapy. Secondary endpoints include: 1) demonstration of stability or improvement in parameters of copper metabolism; 2) improvement in adherence to therapy; 3) no progression of liver disease (defined by changes in synthetic function, albumin and INR, and fibrosis by Fibrotest).

DETAILED DESCRIPTION:
Wilson disease is a genetic disorder of copper metabolism inherited in an autosomal recessive fashion that afflicts ~1/30,000 individuals. Treatment for these individuals consists of medical therapy, which is life-long, or liver transplantation. Medical therapy utilizes chelating agents, penicillamine and trientine, or zinc, each given in multiple daily dosages (1). It is estimated that ~10-50% of individuals have some period of non-adherence to their therapy during their life-time. The consequences of non-adherence include liver injury, liver failure, neurological impairment and death. Some non-adherent individuals can be rescued by reinstitution of medical therapy, while others require liver transplantation (1-4). In addition to the human suffering engendered by the advance in an individuals disease suffered from non-adherence, the physical or mental disability suffered or the need for liver transplantation adds greatly to their cost of life-time care. Simplifying the current treatment regimen for long-term maintenance therapy for Wilson disease should improve patient adherence. This will translate into a positive long-term benefit for patients, their caregivers and supports, and for society as a whole.

Current maintenance therapy for Wilson disease includes the chelating agents penicillamine and trientine, or zinc. Multiple daily dosages (three or four) are recommended from early studies on these medications, by the manufacturer and by treating physicians (1,5-8). As noted above, patient adherence to treatment, and in particular to multiple daily dosages is often incomplete. There has been an increase in the treatment of other common disorders with medication that can be administered as a single daily dosage. As an example, some anti-hypertensives and antidepressants are available in extended release formulations, making a single daily dosage possible. None of the currently available agents for the treatment of Wilson disease has a comparable formulation. Furthermore, even if an extended release oral formulation were available, it is not certain that it would be effective. In an extended release formulation, the site of absorption of the medication may not be sustained adequately, and binding to ingested food may interfere with its function.

The choice of trientine as the single agent for use for study comes from personal experience of the Principal Investigator with its' use in the clinical setting and in a clinical trial (1, 9). This drug has an excellent safety profile and is effective in removing copper from the body when given apart from meals (1,4,10). Previous studies have shown the effectiveness of copper removal by administration in multiple daily dosages (10,11). The amount of copper excreted in the urine of patients on a daily basis is dosage dependent, and is also dependent on the phase of treatment. In the initial treatment period, there is a larger efflux of copper in the urine of patients treated with chelation agents, and with time this amount decreases. For example, patients maintained on d-penicillamine initially may excrete over one milligram of copper in a 24 hour period, but over time will excrete ~250 mcg copper per day. Similarly, patients maintained on trientine as a single therapy may excrete slightly less but comparable amounts of copper (11). In the trials of trientine for neurological disease, the amount of free serum copper and urine copper was stable by the end of the initial 8 week period in most patients (9). Once equilibrium is achieved with respect to copper balance and liver function is stabilized, maintenance therapy is geared towards a smaller net negative removal of copper on a daily basis. Therefore, adequate copper removal should be possible to achieve with an appropriate dosage of trientine given once daily since there is known to be a dose response between trientine and copper excretion.

Supportive evidence suggesting that the single daily dosage proposed in this study will be effective therapy was recently obtained by review of three individual case studies. These three patients, two followed by the principal investigator (MLS) and the third known to him but followed locally, reported taking their trientine as a single daily dosage. Two of the patients had presented with neurological Wilson disease, while the third was a presymptomatic patient identified by family screening; all were years out from their initial treatment. Two of the three changed their regimens to once a day treatment on their own without the advice of their physician due to difficulty taking multiple dosages during their working hours or interference with taking other medications, and the third did so at the advice of another physician. Each of these patients had used single dose therapy for years (range 2-15). Laboratory data for these individuals demonstrated normal liver function and good copper control, and examinations showed them to be clinically stable. All three had previously been treated with d- Penicillamine and then trientine in multiple daily dosages.

Experimental Design & Methods:

Experimental design: Patients meeting inclusion criteria will be asked for their consent to participate in this study before entry into the clinical trial. Patients will be evaluated prior to the start of the study by the Principal Investigator or a co-investigator to document the medical history and physical exam findings. Initial lab studies will be performed to determine the current status of the patient's liver disease and copper balance. A history will be obtained about treatment for their Wilson disease, and patients will be asked to complete a pre-study questionnaire.

Blood and urine studies prior to entry will include: CBC with platelets; Liver function panel (AST, ALT, alkaline phosphatase, total bilirubin, direct bilirubin, GGPT, albumin), INR, serum copper, serum ceruloplasmin, ANA with titer, ESR, pregnancy test, 24 hour urine for copper and zinc and volume, urinalysis and a non-invasive test for liver fibrosis (Fibrotest, Prometheus) A questionnaire will be administered prior to entry into this study and at the end of the study period. This questionnaire is designed to focus on a patients use of their current medications, and at the end of the period, to determine whether the once a day regimen was a useful intervention for them.

For the first part of the study (3 months), the patient will be observed on their current therapy with labs performed prior to study entry and monthly for baseline measurements of liver function and copper status. Subsequently, and throughout the remainder of the study period, patients will be given Trientine at a dosage of ~15 mg/kg rounded upwards to the nearest 250 or 300 mg in a single daily dosage. The entire daily dosage will be taken at once in the AM an hour before any meal. Patients will be monitored monthly for the first three months, and thereafter, every third month by repeat blood and urine testing as noted above, with the exception of the Fibrotest, ANA and ESR that will be administered before the study drug is given, and 12 months later. This interval of monitoring exceeds the frequency at which patients are normally seen for their maintenance therapy, which varies from 3-6 month intervals with the upper limit for those patients with good adherence to past therapy. Patients will be examined at the beginning of the trial, after 3 months after being given study drug, and again after 6 and 12 months of treatment (end of the trial). A monthly study log will be kept by the patient to record their medication administration and any adverse effects of their treatment, and will be sent to the study coordinator.

For long-term follow-up, patients may visit with Dr. Schilsky in our clinic at 6 month intervals for up to ten years (the routine interval for follow-up care for most patients with Wilson disease on maintenance therapy) and standard of care lab testing will be performed. The patient will be asked to fill out a short questionnaire, and data from this visit will be collected and recorded on the case report form. If a patient is unable to travel to the study site, the questionnaire can be filled out by telephone interview and laboratory requests may be sent to the patient for them to have testing and physical examination done locally. Results of these tests and evaluation will be forwarded to our site for review and for data entry.

The study pharmacy will dispense medications at the visit after the third month of monitoring (prior to the initial start of the medication), and thereafter at 90 day intervals. All unused medication will be returned to the study pharmacy.

Methodology Study Group: Patients with an established diagnosis of Wilson disease that have been treated for their disease for at least one year, compensated liver disease and/or stable neurological or psychiatric disease. Biochemical testing must demonstrate normal or minimal elevation of serum ALT (<2 times the upper limit of normal) and a non-ceruloplasmin copper < 25 mcg/dl. Patients must be willing to participate for a 15 month time period and undergo initial monthly blood and urine testing to determine their baseline on their current therapy, and then interval testing for up to 12 months. A pilot study of 5 patients is proposed, with a larger study to follow pending review of the initial pilot data.

ELIGIBILITY:
Inclusion Criteria:

Established diagnosis of Wilson Disease:

* That have been treated for at least 1 year
* Compensated liver disease and/or stable neurological or psychiatric disease.
* Normal or minimal elevation of serum ALT (<2 times upper limit of normal)
* Non-ceruloplasmin copper <25 mcg/dl

Exclusion Criteria:

* Wilson disease diagnosis not well established Wilson disease treated for less than one year Decompensated liver disease (ascites, jaundice, encephalopathy, bleeding due to portal hypertension) Liver disease with elevations of ALT > 2 times upper limit of normal A female who is pregnant or intends to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schilsky, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Background] Roberts EA, Schilsky ML; Division of Gastroenterology and Nutrition, Hospital for Sick Children, Toronto, Ontario, Canada. A practice guideline on Wilson disease. Hepatology. 2003 Jun;37(6):1475-92. doi: 10.1053/jhep.2003.50252. No abstract available. PMID 12774027
- [Background] Schilsky ML, Scheinberg IH, Sternlieb I. Liver transplantation for Wilson's disease: indications and outcome. Hepatology. 1994 Mar;19(3):583-7. doi: 10.1002/hep.1840190307. PMID 8119682
- [Background] Emre S, Atillasoy EO, Ozdemir S, Schilsky M, Rathna Varma CV, Thung SN, Sternlieb I, Guy SR, Sheiner PA, Schwartz ME, Miller CM. Orthotopic liver transplantation for Wilson's disease: a single-center experience. Transplantation. 2001 Oct 15;72(7):1232-6. doi: 10.1097/00007890-200110150-00008. PMID 11602847
- [Background] Askari FK, Greenson J, Dick RD, Johnson VD, Brewer GJ. Treatment of Wilson's disease with zinc. XVIII. Initial treatment of the hepatic decompensation presentation with trientine and zinc. J Lab Clin Med. 2003 Dec;142(6):385-90. doi: 10.1016/S0022-2143(03)00157-4. PMID 14713890
- [Background] Brewer GJ, Dick RD, Johnson VD, Fink JK, Kluin KJ, Daniels S. Treatment of Wilson's disease with zinc XVI: treatment during the pediatric years. J Lab Clin Med. 2001 Mar;137(3):191-8. doi: 10.1067/mlc.2001.113037. PMID 11241029
- [Background] Ferenci P. Wilson's Disease. Clin Gastroenterol Hepatol. 2005 Aug;3(8):726-33. doi: 10.1016/s1542-3565(05)00484-2. PMID 16233999
- [Background] Brewer GJ, Askari F, Lorincz MT, Carlson M, Schilsky M, Kluin KJ, Hedera P, Moretti P, Fink JK, Tankanow R, Dick RB, Sitterly J. Treatment of Wilson disease with ammonium tetrathiomolybdate: IV. Comparison of tetrathiomolybdate and trientine in a double-blind study of treatment of the neurologic presentation of Wilson disease. Arch Neurol. 2006 Apr;63(4):521-7. doi: 10.1001/archneur.63.4.521. PMID 16606763
- [Background] Scheinberg IH, Jaffe ME, Sternlieb I. The use of trientine in preventing the effects of interrupting penicillamine therapy in Wilson's disease. N Engl J Med. 1987 Jul 23;317(4):209-13. doi: 10.1056/NEJM198707233170405. PMID 3600712
- [Background] Walshe JM. Treatment of Wilson's disease with trientine (triethylene tetramine) dihydrochloride. Lancet. 1982 Mar 20;1(8273):643-7. doi: 10.1016/s0140-6736(82)92201-2. PMID 6121964
- [Background] Ferenci P, Caca K, Loudianos G, Mieli-Vergani G, Tanner S, Sternlieb I, Schilsky M, Cox D, Berr F. Diagnosis and phenotypic classification of Wilson disease. Liver Int. 2003 Jun;23(3):139-42. doi: 10.1034/j.1600-0676.2003.00824.x. PMID 12955875
- [Derived] Ala A, Aliu E, Schilsky ML. Prospective pilot study of a single daily dosage of trientine for the treatment of Wilson disease. Dig Dis Sci. 2015 May;60(5):1433-9. doi: 10.1007/s10620-014-3495-6. Epub 2015 Jan 21. PMID 25605552

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Once a Day Trientine
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Once a Day Trientine
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8
Prior Treatment [Number; unit: participants] — Treatment for Wilson's Disease prior to study entry
  participants
    zinc acetate | 2
    d-penicillamine | 1
    trientine BID | 5

OUTCOME MEASURES:

1. Primary Outcome: ALT
Description: Alanine transaminase
Time Frame: Pre Treatment (mean)
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Once a Day Trientine
Number analyzed (Participants) | 8
U/L | 41.38 (31.81)

2. Primary Outcome: ALT
Description: Alanine transaminase
Time Frame: Months 1,2,3,6,9,12 (mean)
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Once a Day Trientine
Number analyzed (Participants) | 8
U/L | 50.89 (32.29)

3. Secondary Outcome: INR
Description: The International Normalized Ratio (INR) is a standard way to describe the time it takes for blood to clot; an INR range of 0.8 to 1.2 is considered normal for a healthy person who is not using oral anticoagulant therapy
Time Frame: Pre Treatment (mean)
Measure: Mean (Standard Deviation); unit: international normalized ratio
Arm/Group | Once a Day Trientine
Number analyzed (Participants) | 8
international normalized ratio | 0.99 (0.07)

4. Secondary Outcome: INR
Description: as for outcome 3
Time Frame: Months 1,2,3,6,9,12 (mean)
Measure: Mean (Standard Deviation); unit: international normalized ratio
Arm/Group | Once a Day Trientine
Number analyzed (Participants) | 8
international normalized ratio | 1.05 (0.08)

5. Secondary Outcome: Albumin
Time Frame: Pre Treatment (mean)
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Once a Day Trientine
Number analyzed (Participants) | 8
g/dL | 0.54 (0.30)

6. Secondary Outcome: Albumin
Time Frame: Months 1,2,3,6,9,12 (mean)
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Once a Day Trientine
Number analyzed (Participants) | 8
g/dL | 0.52 (0.30)

7. Primary Outcome: Cu Serum
Time Frame: Pre Treatment (mean)
Measure: Mean (Standard Deviation); unit: mcg/24h
Arm/Group | Once a Day Trientine
Number analyzed (Participants) | 8
mcg/24h | 0.54 (0.30)

8. Primary Outcome: Cu Serum
Time Frame: Months 1,2,3,6,9,12 (mean)
Measure: Mean (Standard Deviation); unit: mcg/24h
Arm/Group | Once a Day Trientine
Number analyzed (Participants) | 8
mcg/24h | 0.52 (0.30)

9. Secondary Outcome: Cu Urine
Time Frame: Pre Treatment (mean)
Measure: Mean (Standard Deviation); unit: mcg/24hr
Arm/Group | Once a Day Trientine
Number analyzed (Participants) | 8
mcg/24hr | 287.9 (259.1)

10. Secondary Outcome: Cu Urine
Time Frame: Months 1,2,3,6,9,12 (mean)
Measure: Mean (Standard Deviation); unit: mcg/24hr
Arm/Group | Once a Day Trientine
Number analyzed (Participants) | 8
mcg/24hr | 313.4 (191.7)

11. Secondary Outcome: Zn Urine
Time Frame: Pre Treatment (mean)
Measure: Mean (Standard Deviation); unit: mcg/24hr
Arm/Group | Once a Day Trientine
Number analyzed (Participants) | 8
mcg/24hr | 1959 (2214)

12. Secondary Outcome: Zn Urine
Time Frame: Months 1,2,3,6,9,12 (mean)
Measure: Mean (Standard Deviation); unit: mcg/24hr
Arm/Group | Once a Day Trientine
Number analyzed (Participants) | 8
mcg/24hr | 2214 (1346)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Once a Day Trientine
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No